CLINICAL TRIAL: NCT03994107
Title: A Single-center, Prospective, Single Arm Study of Neoadjuvant Treatment With Pegylated Liposomal Doxorubicin（PLD）Plus Albumin-Bound Paclitaxel and Trastuzumab in HER-2 Positive Breast Cancer
Brief Title: Pegylated Liposomal Doxorubicin Plus Albumin-Bound Paclitaxel and Trastuzumab in HER-2 Positive Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Fei Ma, Principal Investigator, Peking Union Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DMS-BC-17
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Albumin-Bound Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLD/albumin-bound paclitaxel/Trastuzumab (Experimental): First phase
  PLD: Level 1：30mg/m2； Level 2：35mg/m2； Level 3：40mg/m2； IV, d1, q21d×6.
  albumin-bound paclitaxel: 220mg/m2 IV for the first infusion，Subsequent infusions 260mg/m2,if no serious adverse reactions occur. d1, q21d×6.
  Trastuzumab：8mg/kg IV for the first infusion , Subsequent infusions 6mg/kg. d1, q21d×6.
  Second phase
  PLD: maximum tolerated dose (MTD). IV, d1, q21d×6.
  albumin-bound paclitaxel: 220mg/m2 IV for the first infusion，Subsequent infusions 260mg/m2,if no serious adverse reactions occur. d1, q21d×6.
  Trastuzumab：8mg/kg IV for the first infusion ,Subsequent infusions 6mg/kg. d1, q21d×6.
  Interventions: Drug: Pegylated Liposomal Doxorubicin; Drug: Albumin-bound paclitaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicin — First phase PLD: 30mg/m2；35mg/m2；40mg/m2；IV, d1, q21d×6.
  Second phase
  PLD：MTD. IV, d1, q21d×6.
Drug: Albumin-bound paclitaxel — 220mg/m2 IV for the first infusion，Subsequent infusions 260mg/m2,if no serious adverse reactions occur. d1, q21d×6.
Drug: Trastuzumab — 8mg/kg IV for the first infusion. Subsequent infusions 6mg/kg. d1, q21d×6.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pegylated liposomal doxorubicin（PLD）plus Albumin-Bound Paclitaxel and trastuzumab as neoadjuvant therapy in HER-2 positive breast cancer.

DETAILED DESCRIPTION:
This is a single-center, prospective, single arm phase II study. Eligible patients will receive neoadjuvant therapy with pegylated liposome doxorubicin (PLD)/albumin-bound paclitaxel/trastuzumab regimentation.

This study consists of two phases, the first phase aims to determine the maximum tolerated dose (MTD) of PLD, and the second phase will explore the efficacy and safety of the regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and voluntarily receive the research procedures according to protocol,willingness to sign the written informed consent document;
2. Female patients aged from 18 to 70 years old;
3. Histologically confirmed as invasive breast cancer. occult breast cancer, inflammatory breast cancer and eczematoid carcinoma are ineligible;
4. Clinical stageⅡ-Ⅲ;
5. HER-2 Positive（defined by: IHC 3+ or ISH positive）;
6. Without previous treatment for this breast cancer;
7. Patients must have at least one measurable disease according to RECIST 1.1;
8. ECOG (Eastern Cooperative Oncology Group) performance score of 0-1 points;
9. LVEF≥55%;
10. Normal ECG;
11. Bone marrow function:absolute neutrophil count (ANC)≥2.0×109/L，platelets≥100×109/L，hemoglobin ≥90g/L。
12. Hepatic function：alanine aminotransferase(ALT) and aspartate aminotransferase(AST) ≤1.5×ULN，serum total bilirubin≤ ULN;
13. Renal function：serum creatinine≤1.5×ULN； Coagulation function：the international standardized ratio (INR) ≤1.5×ULN, prothrombin time (PT) or the activated partial thrombin time (APTT) ≤1.5×ULN.

Exclusion Criteria:

1. New York Heart Association (NYHA) class ≥Ⅱ heart failure.
2. Known or suspected hypersusceptibility to any agents used in the treatment protocol.
3. Need to Concurrent treatment with any other anti-cancer therapy considered by the investigator.
4. participating in other clinical trials within 4 weeks before this study.
5. Serious heart disease, including but not limited to:

1) Significant ventricular arrhythmia or high degree atrioventricular block (Mobitz II or third degree atrioventricular block); 2) unstable angina; 3) clinically significant heart valve disease; 4) Electrocardiogram shows transmural myocardial infarction; 5) Uncontrolled hypertension. 6. Uncontrolled diabetes. 7. Severe or uncontrolled infection. 8. Hepatitis b surface antigen positive, or hepatitis c virus antibody positive, or human immunodeficiency virus (HIV) antibody positive.

9. Active malignancy, other than adequately treated carcinoma in situ of the cervix or basal cell carcinoma of the skin，within the past 5 years.

9）Women who are pregnant , breastfeeding ,or refuse to use adequate contraception prior to study entry and for the duration of study participation.

10）Other conditions considered to be inappropriate to be enrolled by the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response(pCR) rate | 5 months
  Percentage of patients who do not exhibit residual invasive breast cancer in breast and lymph nodes at time of surgery

SECONDARY OUTCOMES:
Rate of Breast conserving surgery | 5 months
  Percentage of patients undergoing breast-conserving surgery after neoadjuvant therapy
Rate of surgery | 5 months
  Percentage of patients undergoing mastectomy and breast-conserving surgery after neoadjuvant therapy
adverse events | 5 months
  Incidence and Severity of adverse events ,according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ma, MD, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (1):
- Fei Ma, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided